CLINICAL TRIAL: NCT05822440
Title: A Phase 1, Open-Label, 2-Period, Fixed Sequence Study to Estimate the Effect of Itraconazole on the Pharmacokinetics of PF-07817883 in Healthy Adults
Brief Title: A Study to Learn About How Itraconazole Affects the Blood Level of Study Medicine (PF-07817883) in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C5091008
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Itraconazole

STUDY DESIGN:
Masking Description: Masking: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): The treatment arm includes a single dose of PF-07817883 (Period 1 Day 1)
  Interventions: Drug: PF-07817883
- Period 2 (Experimental): This treatment arm includes 7-day dosing of itraconazole with a single dose of PF-07817883 Co-administered on Day 4 (Period 2 Day 4)
  Interventions: Drug: PF-07817883; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-07817883 — Single oral dose (period 1) or co-administered with itraconazole (period 2)
Drug: Itraconazole — Interacting drug which will be given for 7 days in period 2
  Other Names: Sporanox®
  Arms: Period 2

SUMMARY:
The purpose of this study is to learn how Itraconazole affects the blood level of PF-07817883 in Healthy Adults.

This study is seeking participants who are:

* male and female aged 18 to 65 years old,
* overtly healthy. This can be determined my medical evaluation, medical history, lab tests etc.

This study will consist of 2 parts, Period 1 and Period 2.

Period 1: participants will take PF-07817883 one time by mouth at the study clinic.

Period 2: participants will take PF-07817883 one time by mouth at the study clinic. They will also take daily itraconazole by mouth for 7 days.

Participants will stay at the study clinic for 2 weeks in total. The study doctors will collect blood and urine samples from everyone. The study doctors will check participants' reactions to the study medicine for safety measures. There is a follow-up call at 28 to 35 days from the last dose of PF-07817883.

Itraconazole is an approved medicine. It is also a metabolism inhibitor. When taken with some medicines, it affects the actual level of these medicines in the body. This study will compare blood levels of PF-07817883 given with and without Itraconazole. This will help decide safety and right amount for PF-07817883 when given with metabolism inhibitors.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, 2-period, fixed sequence study to estimate the effect of itraconazole, a strong CYP3A4 inhibitor, on the plasma PK of PF-07817883 in healthy adults. The study will consist of 2 treatments: a single oral dose of PF-07817883 alone and a single oral dose of PF-07817883 in combination with multiple oral doses of itraconazole. The PK and safety will be assessed and compared for single dose of PF-07817883 in period 1 and period 2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 65 years of age, inclusive, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and standard 12-lead ECG.
* BMI of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, CV, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Positive test result for SARS-CoV-2 infection at admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants were enrolled in the study. Study had 2 treatment periods with fixed sequence.
Groups:
- PF-07817883: Participants received PF-07817883 300 milligrams (mg) as a single oral dose on Day 1 of Period 1.
- PF-07817883 + Itraconazole: Participants received itraconazole 200 mg orally once in a day (QD) from Day 1 to Day 7 of Period 2. On Day 4 of Period 2, participants received PF-07817883 300 mg as a single oral dose.
Period: Treatment Period 1 (5 Days)
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Treatment Period 2 (8 Days)
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Started | 0 | 12 (Participants entered Period 2.)
Completed | 0 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- All Participants: All participants who received PF-07817883 300 mg orally on Day 1 of Period 1 and on Day 4 of Period 2 along with itraconazole 200 mg QD orally from Day 1 to Day 7 of Period 2.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of PF-07817883
Description: Cmax was observed directly from data and measured in nanogram per milliliter (ng/mL).
Time Frame: Period 1: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose on Day 1; Period 2: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose on Day 4
Population: Pharmacokinetic (PK) parameter set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 11
ng/mL | 4030 (28) | 4985 (41)
Statistical Analysis 1: Comparison: PF-07817883 vs PF-07817883 + Itraconazole; Ratio was between test to reference, where test is PF-07817883 + Itraconazole arm and reference is PF-07817883 arm. Natural log transformed Cmax of PF-07817883 were analyzed using a mixed effect model with treatment as fixed effect and participant as a random effect. The ratios (and 90% CIs) were expressed as percentages; Test type: Other; Ratio of Adjusted Geometric Means = 124.35, 90% CI 2-sided [100.22 to 154.29]

2. Primary Outcome: Area Under the Concentration -Time Curve From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of PF-07817883
Description: AUCinf was derived by AUClast + (Clast*/kel). AUClast was area under the plasma concentration-time profile from time 0 to the time of Clast; Clast* was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve. AUCinf was measured in nanogram*hour per milliliter (ng*hr/mL).
Time Frame: as for outcome 1
Population: PK parameter set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 11
ng*hr/mL | 21720 (26) | 46400 (36)
Statistical Analysis 1: Comparison: PF-07817883 vs PF-07817883 + Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 212.83, 90% CI [183.76 to 246.50]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. TEAEs were events that occurred between first dose of study intervention and up to maximum of 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 of dosing up to 35 days post last dose of study intervention (maximum up to 48 days)
Population: Safety analysis set included all participants enrolled and took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Itraconazole: Participants received itraconazole 200 mg orally once in a day (QD) alone from first dose of itraconazole administered alone in Period 2 Day 1 up to just before coadministration of PF-07817883 in Period 2 Day 4.
- Itraconazole + PF-07817883: Participants received itraconazole 200 mg QD with PF-07817883 300 mg SD from coadministration of PF-07817883 with itraconazole in Period 2 Day 4 through the end of the study.
Arm/Group | PF-07817883 | Itraconazole | Itraconazole + PF-07817883
Number analyzed (Participants) | 12 | 12 | 12
Participants | 1 | 3 | 2

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory assessments included: hematology assessments included monocytes/leukocytes (percentage [%]) greater than (>) 1.2*upper limit of normal (ULN), urinalysis assessments included urine hemoglobin greater than or equal to (>=) 1, low power field (LPF), urine bacteria >20/LPF.
Time Frame: Day 1 of dosing up to last dose of study intervention or early termination/discontinuation (maximum up to 13 days)
Population: Safety analysis set included all participants enrolled and took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 12
Participants | 0 | 3

5. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings Per Pre-defined Criteria
Description: Standard 12-lead ECGs was collected using an ECG system that automatically calculates the heart rate (HR) and measures PR interval, QT interval, QTcF, and QRS interval. All scheduled ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position. To ensure safety of the participants, a qualified individual at the investigator site made comparisons to baseline measurements. Pre-defined criteria was defined as 30 milliseconds (ms) less than (<) change less than or equal to (<=) 60 ms.
Time Frame: Day 1 of dosing up to last dose of study intervention or early termination/discontinuation (maximum up to 13 days)
Population: Safety analysis set included all participants enrolled and took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1

6. Secondary Outcome: Number of Participants With Vital Signs Findings Per Pre-defined Criteria
Description: Vital signs included: supine diastolic blood pressure (DBP) measured in millimetre of mercury (mmHg) with criteria value as follows- Value <50 mmHg, change>= 20 mmHg increase, change >= 20 mmHg decrease; supine pulse rate (PR) measured in beats per minute (bpm) with criteria values as follows- value < 40 bpm, value > 120 bpm; supine systolic blood pressure (SBP, mmHg) with criteria values as follows- value< 90 mmHg, change >= 30 mmHg increase, change >=30 mmHg decrease. Vital signs (SBP BP, and pulse rate) were measured with participants after having a rest for at least 5 minutes in a supine position. Supine BP was measured with the participant's arm supported at the level of the heart and recorded to the nearest mmHg after approximately 5 minutes of rest. If timing of these measurements coincided with a blood collection, BP and PR were obtained prior to nominal time of blood collection. Only participants having at least 1 vital sign findings per pre-defined criteria are reported.
Time Frame: Day 1 of dosing up to last dose of study intervention or early termination/discontinuation (maximum up to 13 days)
Population: Safety analysis set included all participants enrolled and took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: A complete physical examination included, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A brief physical examination included, at a minimum, assessments of general appearance, the respiratory and CV systems, and participant-reported symptoms. Physical examinations were conducted by a physician, trained physician's assistant, or nurse practitioner as acceptable according to local regulation. Clinical significance of physical examination abnormalities was judged by physicians.
Time Frame: Day 1 of dosing up to last dose of study intervention or early termination/discontinuation (maximum up to 13 days)
Population: Safety analysis set included all participants enrolled and took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

8. Secondary Outcome: Time to Reach Cmax (Tmax) of PF-07817883
Description: Tmax is the time taken (in hours) to reach the maximum serum drug concentration. Tmax was observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 11
Hours | 1.76 [0.517 to 4.03] | 2.00 [1.52 to 4.00]

9. Secondary Outcome: Terminal Phase Half-Life (t1/2) of PF-07817883
Description: Terminal half-life was defined as the time measured for the plasma concentration of drug to decrease by one half. t1/2 was determined by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 11
Hours | 5.502 (2.3703) | 10.92 (8.3667)

10. Secondary Outcome: Apparent Clearance (CL/F) of PF-07817883
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as dose administered divided by area under the concentration curve from time 0 extrapolated to infinite time (AUCinf).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/Hours
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 11
Liter/Hours | 13.81 (26) | 6.469 (36)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07817883
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-07817883 | PF-07817883 + Itraconazole
Number analyzed (Participants) | 12 | 11
Liter | 100.4 (63) | 86.29 (51)

ADVERSE EVENTS:
Time Frame: Day 1 up to 35 days after last dose of study drug (maximum up to 48 days)
Arm/Group | PF-07817883 | Itraconazole | Itraconazole + PF-07817883
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07817883 (N=12) | Itraconazole (N=12) | Itraconazole + PF-07817883 (N=12)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05822440/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT05822440/SAP_001.pdf